CLINICAL TRIAL: NCT03777293
Title: Guangdong Key Laboratory of Liver Disease Research, Department of Medical Ultrasound, The Third Affiliated Hospital of Sun Yat-sen University
Brief Title: A Prospective Study to Monitor Liver Diseases Dynamically by Ultrasound Viscoelasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Rongqin Zheng, Guangdong Key Laboratory of Liver Disease Research, Department of Medical Ultrasound, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: sysu2018
Record Dates: First submitted 2018-12-11; First posted 2018-12-17 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Cirrhosis; Liver Diseases
MeSH Terms: conditions — Fibrosis; Liver Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training cohort (Experimental): ultrasound viscoelasticity
  Interventions: Device: ultrasound viscoelasticity
- testing cohort (Other): ultrasound viscoelasticity
  Interventions: Device: ultrasound viscoelasticity

INTERVENTIONS:
Device: ultrasound viscoelasticity — use these devices to do ultrasound examination in chronic liver disease patients
  Other Names: LOGIQ E produced by GE; Aplio i900 produced by Canon

SUMMARY:
The accuracy of ultrasound elastography for assessing liver fibrosis by measuring liver stiffness (elastic modulus) is better than traditional method. Elastography has certain advantage such as non-invasive, simple, real-time and it has been recommended by clinical guidelines.

However, some chanllenging scientific problems showed up with further research and clinical practice. Firstly, present elastography machines can only calculate liver stiffness from shear wave speed or elastic modulus but ignore other physical characteristics such as tissue viscosity. So far, present technique simply assume liver as an idealized model with isotropic elasticity to assess liver fibrosis while liver is actually anisotropic and viscoelastic. What's more, theoretically, there are not only different solid state structures such as cell organization and vessel but also flowing liquid such as blood and bile. Thus, ignoring viscosity and evaluating elasticity only is unreasonable. In the other hand, a number of confounding factors have been found to influence liver stiffness measurement by elastography. Different pathological chang of liver including inflammation, necrosis, cholestasis and inhomogeneity among the individuals such as obesity, ascites, et,al. will decrease the accuracy of liver stiffness measurement and liver fibrosis staging by elastography.

In fact, liver fibrosis is a dynamic process. Liver fibrosis is a reaction of compensation and repair for inflammation and necrosis as well as a contributing factor for liver damage. This dynamic process constitutes the common characteristic of chronic liver disease and result in the complicated biological mechanical characteristics of liver. In consequence, how to measure liver viscosity and elasticity respectively, and to evaluate liver fibrosis stage and Inflammation degree accurately during the complicated and dynamic pathological process is the key scientific problem demanding solution, which is also the urgent requirement of related fundamental research and clinical practice.

Therefore, this project plan to apply LOGIQ E viscoelastography machine as research tool, rat liver fibrosis model and rat liver failure model as research object to investigate the correlation between liver viscoelastography measurement and liver fibrosis stage and Inflammation degree. The investigators also aim to assess the feasibility of using ulstrasound viscoelastography to evaluate liver fibrosis stage and Inflammation degree dynamically.

ELIGIBILITY:
Inclusion Criteria:

* agree to have liver biopsy in later therapy
* agree to participate in our study

Exclusion Criteria:

* Hepatic malignant mass lesion
* After liver transplantation
* Pregnant patients
* Liver biopsy specimens do not meet the requirements: speciments length <15mm, or numbers of the portal ducts <6.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
liver fibrosis stage | 1 year
  the degree of liver fibrosis according to metavir scores.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Rongqin, phd, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The department of Ultrasound, the third affiliated hospital of Sun Yat-son University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang XQ, Zheng RQ, Jin JY, Wang JF, Zhang T, Zeng J. US Shear-Wave Elastography Dispersion for Characterization of Chronic Liver Disease. Radiology. 2022 Dec;305(3):597-605. doi: 10.1148/radiol.212609. Epub 2022 Aug 2. PMID 35916675